CLINICAL TRIAL: NCT03255811
Title: Clinical Study on Treatment of Apatinib Mesylate in First-line Maintenance of Advanced Gastric Cancer -- Multicenter, Open, One Arm Exploratory Study
Brief Title: Clinical Study on Treatment of Apatinib Mesylate in First-line Maintenance of Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: DongMa (Other)
Responsible Party: Sponsor-Investigator, DongMa, Director of gastrointestinal oncology, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gastrointestinal cancer
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced gastric cancer apatinib Maintenance therapy
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Intervention Model Description: At present, apatinib was approved for the treatment of advanced gastric cancer after second-line or gastroesophageal junction adenocarcinoma, is in the second one, experience of medication, clinical data, no chemotherapy so now intends to carry out 40 cases of small sample exploratory research, in the conventional chemotherapy after the onset, with APA for Nigeria maintenance treatment, with a preliminary understanding of apatinib in first-line advanced gastric cancer to maintain the efficacy and safety of the treatment, and explore the feasibility of anti generate small molecule targeted therapy in advanced gastric cancer vascular pattern.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dosage regimen (Experimental): The chemotherapy response rate reached the maximum after 14-28 days, apatinib, 750 mg (QD), once a day, half an hour after meal (daily dosing time should be as same as possible), with warm boiling water delivery service. 28 days for a dosing cycle.
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — Apatinib mesylate tablets treatment and to maintain the actual benefit in progression free survival.

SUMMARY:
At present, apatinib was approved for the treatment of advanced gastric cancer after second-line or gastroesophageal junction adenocarcinoma, is in the second one, experience of medication, clinical data, no chemotherapy so now intends to carry out 40 cases of small sample exploratory research, in the conventional chemotherapy after the onset, with APA for Nigeria maintenance treatment, with a preliminary understanding of apatinib in first-line advanced gastric cancer to maintain the efficacy and safety of the treatment, and explore the feasibility of anti generate small molecule targeted therapy in advanced gastric cancer vascular pattern.

DETAILED DESCRIPTION:
The incidence of gastric cancer in China is high, and there is no standard first-line chemotherapy regimen for advanced gastric cancer. Second-line therapy usually involves first-line treatment, without the use of drugs for combination or monotherapy, and no uniform treatment. Apatinib approved provides a good solution to this problem, but this study is in limit of validity standard after all into the row, not very good reaction in clinical practice for APA imatinib reality in the treatment of advanced gastric cancer. Therefore, it is necessary to make a prospective product study to understand the gap between clinical practice and research results. This study can evaluate apatinib in treatment of advanced gastric or gastroesophageal junction safe and effective parts of adenocarcinoma in clinical practice, and the specific usage (such as dose and period). The results of this study can help the future clinical practice specification of apatinib parts for the treatment of adenocarcinoma with advanced gastric or gastroesophageal reflux, the advanced gastric or gastroesophageal adenocarcinoma patients with parts get treatment more safe and effective in the treatment of.

At present, apatinib was approved for the treatment of advanced gastric cancer after second-line or gastroesophageal junction adenocarcinoma, is in the second one, experience of medication, clinical data, no chemotherapy so now intends to carry out 40 cases of small sample exploratory research, in the conventional chemotherapy after the onset, with APA for Nigeria maintenance treatment, with a preliminary understanding of apatinib in first-line advanced gastric cancer to maintain the efficacy and safety of the treatment, and explore the feasibility of anti generate small molecule targeted therapy in advanced gastric cancer vascular pattern.

ELIGIBILITY:
Inclusion Criteria:

1. age: more than 18 years old, male or female;
2. histologically confirmed advanced gastric or gastroesophageal junction adenocarcinoma, stomach with measurable lesions (spiral CT scan is more than 10mm, meet the RECIST standard 1.1);
3. inoperable, locally advanced, recurrent or metastatic adenocarcinoma of the stomach or esophagogastric junction;
4. first-line chemotherapy (oxaliplatin / cisplatin / paclitaxel combined with fluorouracil / either drug, docetaxel or S-1 / capecitabine), efficacy evaluation of SD or CR or PR may, from the last chemotherapy cycle time is not more than 28 days;
5. when evaluating the maximum response rate of chemotherapy (chemotherapy is not less than 4 cycles), enter maintenance therapy. (maximum response rate: compared with the previous curative effect evaluation, the target lesion no longer continued to shrink);
6. ECOG PS:0-1 points;
7. baseline blood routine and biochemical parameters met the following criteria: Hemoglobin is larger than 80g/L,

   * the absolute neutrophil count (ANC) = 1.5 * 109/L, Over 90 * 109/L platelets,
   * ALT, AST less than 2.5 times the upper limit of normal value, Equal to or less than 5 times the upper limit of normal (liver metastasis),
   * the serum total bilirubin is less than 1.5 times the upper limit of normal value, Serum creatinine. Less than 1.5 times the upper limit of normal value, Serum albumin is more than 30g/L;
8. more than the expected survival time in March;
9. women of childbearing age must have pregnancy tests (serum or urine) within 7 days prior to admission, and the results are negative and are willing to take the appropriate method of contraception at 8 weeks after the trial and at the end of the test. For men, surgical sterilization should be applied, or consent to the appropriate method of contraception 8 weeks after the trial and at the end of the trial;
10. subjects voluntarily joined the study, signed informed consent, good compliance, and followed up.

Exclusion Criteria:

1. confirmed of apatinib and / or its accessories allergy;
2. with high blood pressure and the antihypertensive drug treatment can not be reduced to the normal range (>140 systolic blood pressure mmHg, diastolic blood pressure >90 mmHg), with I level above grade I coronary heart disease, arrhythmia (including QTc prolongation > 450 male MS, female MS > 470) and grade I heart function insufficiency; patients with positive urinary protein;
3. , there are a variety of factors that affect oral medication (such as inability to swallow, nausea, vomiting, chronic diarrhea, and intestinal obstruction); The 4. has a clear tendency in patients with gastrointestinal bleeding, including the following: local active ulcerative lesions, and fecal occult blood (+ +) can not be enrolled; 2 months melena, hematemesis history; for fecal occult blood (+) and gastric primary tumor without surgical resection. And for gastroscopy, such as gastric cancer, and researchers believe that may occur in massive hemorrhage of digestive tract were;

5. coagulation dysfunction (INR>1.5, APTT>1.5, ULN), with bleeding tendency; 6. patients with central nervous system metastasis; 7. pregnant or lactating women; A patient with other malignancies within 8.5 years; 9. patients who have history of psychotropic substance abuse and are unable to quit or have mental disorders; Patients who participated in other clinical trials within 10.4 weeks; 11. received VEGFR inhibitors, such as Sola Fini and sunitinib therapy; 12. according to the researcher's judgment, there are patients who seriously endanger the safety of patients or affect the patients who complete the study; 13., the researchers considered unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-01-25 (Estimated); Study Completion 2019-03-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of apatinib mesylate tablets as first-line maintenance treatment for advanced gastric or gastroesophageal junction progression free survival site adenocarcinoma | 2 years
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ma Dong, graduate, Study Director — Leading Investigator
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China